CLINICAL TRIAL: NCT00870012
Title: Treatment of Nonalcoholic Fatty Liver Disease With Probiotics and Prebiotics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Henry LY Chan, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: NAFLD-GUT#2
Record Dates: First submitted 2009-03-25; First posted 2009-03-26 (Estimated); Last update posted 2014-02-24 (Estimated); Status verified 2014-02

CONDITIONS: Nonalcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lepicol probiotic & prebiotic formula+simple lifestyle advice (Active Comparator)
  Interventions: Drug: Lepicol probiotic & prebiotic formula; Other: Simple lifestyle advice
- Simple lifestyle advice alone (Placebo Comparator)
  Interventions: Other: Simple lifestyle advice

INTERVENTIONS:
Drug: Lepicol probiotic & prebiotic formula — NAFLD patients treated with Lepicol probiotic and prebiotic formula for 24 weeks.
  Arms: Lepicol probiotic & prebiotic formula+simple lifestyle advice
Other: Simple lifestyle advice — NAFLD patients treated with lifestyle advice.

SUMMARY:
The investigators' aim is to determine whether probiotic and prebiotic treatment plus lifestyle advice is more effective in reducing hepatic fat content than lifestyle advice alone in patients with Nonalcoholic Fatty Liver Disease (NAFLD).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 70 years
* Fatty liver identified by imaging studies including ultrasound, computer tomography or magnetic resonance imaging
* Elevated alanine aminotransferase (ALT) according to Prati's criteria (>30 IU/l in men and >19 IU/l in women)18
* Written informed consent obtained

Exclusion Criteria:

* Positive hepatitis B surface antigen, anti-hepatitis C virus antibody, or anti-nuclear antibody titer above 1/160
* Alcohol consumption above 30 g per week in men or 20 g per week in women
* ALT above 10 times the upper limit of normal
* Liver decompensation, as evidenced by bilirubin above 50 µmol/l, platelet count below 100 × 109/l, prothrombin time above 1.3 times the upper limit of normal, albumin below 35 g/l, presence of ascites or varices
* Use of systemic corticosteroids and methotrexate in the last 6 months
* Evidence of hepatocellular carcinoma
* Terminal illness or cancer, unless in complete remission for more than 5 years

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-02; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the reduction in hepatic triglyceride content from baseline to week 24. | 24 weeks

SECONDARY OUTCOMES:
The proportion of patients with normal ALT at week 24 will be determined. Normal ALT is defined according to Prati's cutoffs (≤30 IU/l in men and ≤19 IU/l in women). | 24 weeks
The proportion of patients with impaired fasting glucose, diabetes, insulin resistance (estimated by the homeostasis model), hypertension, dyslipidemia and metabolic syndrome will be determined both at baseline and during each visit. | 24 weeks
The changes in visceral fat will be determined by magnetic resonance imaging at the same session both at baseline and month 12. | 12 months
The changes in liver fibrosis will be determined by transient elastography by Fibroscan both at baseline and month 12. | 12 months
The percentage of total sequences of individual microbes will be calculated. In particular, the proportion of Firmicutes and Bacteroidetes will be compared between the two treatment arms. | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Cheng Suen Man Shook Hepatitis Center, Institute of Digestive Disease, The Chinese University of Hong Kong, Prince of Wales Hospital, Hong Kong SAR, China

REFERENCES:
- [Background] Farrell GC, Larter CZ. Nonalcoholic fatty liver disease: from steatosis to cirrhosis. Hepatology. 2006 Feb;43(2 Suppl 1):S99-S112. doi: 10.1002/hep.20973. PMID 16447287
- [Background] Bugianesi E, Leone N, Vanni E, Marchesini G, Brunello F, Carucci P, Musso A, De Paolis P, Capussotti L, Salizzoni M, Rizzetto M. Expanding the natural history of nonalcoholic steatohepatitis: from cryptogenic cirrhosis to hepatocellular carcinoma. Gastroenterology. 2002 Jul;123(1):134-40. doi: 10.1053/gast.2002.34168. PMID 12105842
- [Background] Fassio E, Alvarez E, Dominguez N, Landeira G, Longo C. Natural history of nonalcoholic steatohepatitis: a longitudinal study of repeat liver biopsies. Hepatology. 2004 Oct;40(4):820-6. doi: 10.1002/hep.20410. PMID 15382171
- [Background] Hui AY, Wong VW, Chan HL, Liew CT, Chan JL, Chan FK, Sung JJ. Histological progression of non-alcoholic fatty liver disease in Chinese patients. Aliment Pharmacol Ther. 2005 Feb 15;21(4):407-13. doi: 10.1111/j.1365-2036.2005.02334.x. PMID 15709991
- [Background] Villanova N, Moscatiello S, Ramilli S, Bugianesi E, Magalotti D, Vanni E, Zoli M, Marchesini G. Endothelial dysfunction and cardiovascular risk profile in nonalcoholic fatty liver disease. Hepatology. 2005 Aug;42(2):473-80. doi: 10.1002/hep.20781. PMID 15981216
- [Background] Wong VW, Hui AY, Tsang SW, Chan JL, Tse AM, Chan KF, So WY, Cheng AY, Ng WF, Wong GL, Sung JJ, Chan HL. Metabolic and adipokine profile of Chinese patients with nonalcoholic fatty liver disease. Clin Gastroenterol Hepatol. 2006 Sep;4(9):1154-61. doi: 10.1016/j.cgh.2006.06.011. Epub 2006 Aug 14. PMID 16904946
- [Background] Targher G, Bertolini L, Rodella S, Tessari R, Zenari L, Lippi G, Arcaro G. Nonalcoholic fatty liver disease is independently associated with an increased incidence of cardiovascular events in type 2 diabetic patients. Diabetes Care. 2007 Aug;30(8):2119-21. doi: 10.2337/dc07-0349. Epub 2007 May 22. No abstract available. PMID 17519430
- [Background] Belfort R, Harrison SA, Brown K, Darland C, Finch J, Hardies J, Balas B, Gastaldelli A, Tio F, Pulcini J, Berria R, Ma JZ, Dwivedi S, Havranek R, Fincke C, DeFronzo R, Bannayan GA, Schenker S, Cusi K. A placebo-controlled trial of pioglitazone in subjects with nonalcoholic steatohepatitis. N Engl J Med. 2006 Nov 30;355(22):2297-307. doi: 10.1056/NEJMoa060326. PMID 17135584
- [Background] Lutchman G, Modi A, Kleiner DE, Promrat K, Heller T, Ghany M, Borg B, Loomba R, Liang TJ, Premkumar A, Hoofnagle JH. The effects of discontinuing pioglitazone in patients with nonalcoholic steatohepatitis. Hepatology. 2007 Aug;46(2):424-9. doi: 10.1002/hep.21661. PMID 17559148
- [Background] Balas B, Belfort R, Harrison SA, Darland C, Finch J, Schenker S, Gastaldelli A, Cusi K. Pioglitazone treatment increases whole body fat but not total body water in patients with non-alcoholic steatohepatitis. J Hepatol. 2007 Oct;47(4):565-70. doi: 10.1016/j.jhep.2007.04.013. Epub 2007 May 24. PMID 17560678
- [Background] Samaha FF, Iqbal N, Seshadri P, Chicano KL, Daily DA, McGrory J, Williams T, Williams M, Gracely EJ, Stern L. A low-carbohydrate as compared with a low-fat diet in severe obesity. N Engl J Med. 2003 May 22;348(21):2074-81. doi: 10.1056/NEJMoa022637. PMID 12761364
- [Background] Ley RE, Turnbaugh PJ, Klein S, Gordon JI. Microbial ecology: human gut microbes associated with obesity. Nature. 2006 Dec 21;444(7122):1022-3. doi: 10.1038/4441022a. PMID 17183309
- [Background] Backhed F, Ding H, Wang T, Hooper LV, Koh GY, Nagy A, Semenkovich CF, Gordon JI. The gut microbiota as an environmental factor that regulates fat storage. Proc Natl Acad Sci U S A. 2004 Nov 2;101(44):15718-23. doi: 10.1073/pnas.0407076101. Epub 2004 Oct 25. PMID 15505215
- [Background] Ley RE, Backhed F, Turnbaugh P, Lozupone CA, Knight RD, Gordon JI. Obesity alters gut microbial ecology. Proc Natl Acad Sci U S A. 2005 Aug 2;102(31):11070-5. doi: 10.1073/pnas.0504978102. Epub 2005 Jul 20. PMID 16033867
- [Background] Turnbaugh PJ, Ley RE, Mahowald MA, Magrini V, Mardis ER, Gordon JI. An obesity-associated gut microbiome with increased capacity for energy harvest. Nature. 2006 Dec 21;444(7122):1027-31. doi: 10.1038/nature05414. PMID 17183312
- [Background] Lichtman SN, Sartor RB, Keku J, Schwab JH. Hepatic inflammation in rats with experimental small intestinal bacterial overgrowth. Gastroenterology. 1990 Feb;98(2):414-23. doi: 10.1016/0016-5085(90)90833-m. PMID 2295397
- [Background] Bigorgne AE, Bouchet-Delbos L, Naveau S, Dagher I, Prevot S, Durand-Gasselin I, Couderc J, Valet P, Emilie D, Perlemuter G. Obesity-induced lymphocyte hyperresponsiveness to chemokines: a new mechanism of Fatty liver inflammation in obese mice. Gastroenterology. 2008 May;134(5):1459-69. doi: 10.1053/j.gastro.2008.02.055. Epub 2008 Mar 4. PMID 18471520
- [Background] Prati D, Taioli E, Zanella A, Della Torre E, Butelli S, Del Vecchio E, Vianello L, Zanuso F, Mozzi F, Milani S, Conte D, Colombo M, Sirchia G. Updated definitions of healthy ranges for serum alanine aminotransferase levels. Ann Intern Med. 2002 Jul 2;137(1):1-10. doi: 10.7326/0003-4819-137-1-200207020-00006. PMID 12093239
- [Background] Canani RB, Cirillo P, Terrin G, Cesarano L, Spagnuolo MI, De Vincenzo A, Albano F, Passariello A, De Marco G, Manguso F, Guarino A. Probiotics for treatment of acute diarrhoea in children: randomised clinical trial of five different preparations. BMJ. 2007 Aug 18;335(7615):340. doi: 10.1136/bmj.39272.581736.55. Epub 2007 Aug 9. PMID 17690340
- [Background] Hickson M, D'Souza AL, Muthu N, Rogers TR, Want S, Rajkumar C, Bulpitt CJ. Use of probiotic Lactobacillus preparation to prevent diarrhoea associated with antibiotics: randomised double blind placebo controlled trial. BMJ. 2007 Jul 14;335(7610):80. doi: 10.1136/bmj.39231.599815.55. Epub 2007 Jun 29. PMID 17604300
- [Background] Altschul SF, Madden TL, Schaffer AA, Zhang J, Zhang Z, Miller W, Lipman DJ. Gapped BLAST and PSI-BLAST: a new generation of protein database search programs. Nucleic Acids Res. 1997 Sep 1;25(17):3389-402. doi: 10.1093/nar/25.17.3389. PMID 9254694
- [Background] Cole JR, Chai B, Farris RJ, Wang Q, Kulam SA, McGarrell DM, Garrity GM, Tiedje JM. The Ribosomal Database Project (RDP-II): sequences and tools for high-throughput rRNA analysis. Nucleic Acids Res. 2005 Jan 1;33(Database issue):D294-6. doi: 10.1093/nar/gki038. PMID 15608200
- [Background] Eckburg PB, Bik EM, Bernstein CN, Purdom E, Dethlefsen L, Sargent M, Gill SR, Nelson KE, Relman DA. Diversity of the human intestinal microbial flora. Science. 2005 Jun 10;308(5728):1635-8. doi: 10.1126/science.1110591. Epub 2005 Apr 14. PMID 15831718
- [Derived] Wong VW, Won GL, Chim AM, Chu WC, Yeung DK, Li KC, Chan HL. Treatment of nonalcoholic steatohepatitis with probiotics. A proof-of-concept study. Ann Hepatol. 2013 Mar-Apr;12(2):256-62. PMID 23396737